CLINICAL TRIAL: NCT06107829
Title: Identification, Assessment, and Treatment of Tardive Dyskinesia With Valbenazine in Adults With Intellectual/Developmental Disabilities and Co-occurring Psychiatric and/or Behavioral Disorders
Brief Title: Valbenazine Treatment of Tardive Dyskinesia in Adults With Intellectual/Developmental Disabilities
Acronym: TD-AIDD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not funded
Sponsor: Stephen Ruedrich (Other)
Collaborators: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor-Investigator, Stephen Ruedrich, Physician, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20221555
Record Dates: First submitted 2023-10-25; First posted 2023-10-30 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Tardive Dyskinesia; Intellectual Disability; Developmental Disabilities
Keywords: valbenazine; movement disorders; antipsychotic medication adverse effects; Abnormal Involuntary Movement Scale; quality of life; adaptive behavior; caregiver burden; selective vesicular monoamine transporter 2 inhibitor
MeSH Terms: conditions — Tardive Dyskinesia; Intellectual Disability; Developmental Disabilities; Movement Disorders; Caregiver Burden | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Valbenazine (Experimental): This an open-label study in which all participants will have their valbenazine dose titrated from 40 mg to 80 mg per day, which will remain the valbenazine dose through end of study, unless interrupted by adverse events. Participants taking valbenazine who are concurrently taking strong CYP2D6 inhibitors (paroxetine, fluoxetine, bupropion, duloxetine) will continue their valbenazine dose at 40 mg per day through end of study. Participants taking valbenazine who are concurrently taking strong CYP3A4 inhibitors (ketoconazole, fluconazole, cimetidine, verapamil) will continue their valbenazine dose at 40 mg per day through end of study.
  Interventions: Drug: Valbenazine Oral Capsule

INTERVENTIONS:
Drug: Valbenazine Oral Capsule — Open-label twenty-four-week treatment with valbenazine oral capsules (up to 80 mg/day) to test the safety and effectiveness of this medication in ameliorating the signs of tardive dyskinesia in persons with intellectual disability.
  Other Names: Ingrezza

SUMMARY:
The goal of this open-label clinical trial is to test the safety and efficacy of valbenazine treatment in patients with Intellectual/Developmental Disability (IDD) who have a diagnosis of Tardive dyskinesia (TD). The main questions this study aims to answer are:

* Does valbenazine treatment of TD in the previously untreated patient population of adults with IDD produce comparable amelioration of signs of movement disorder as what has historically been reported in adults without IDD?
* Is valbenazine treatment of TD in persons with IDD as safe as what has historically been reported in adults without IDD?
* Does valbenazine treatment improve Quality of Life (QOL) in persons with IDD and TD treated with valbenazine?
* Does valbenazine treatment produce positive change in Activities of Daily Living (ADLs) in persons with IDD and TD?
* Does valbenazine treatment of TD in persons with IDD reduce caregiver burden?

In this study, 25 participants with IDD and TD will undergo valbenazine treatment for 24 weeks. The participants will be seen for a total of 5 visits: at baseline, and at follow up visits at 3 weeks, 6 weeks, 12 weeks, and 24 weeks.

This study does not include a comparison group. Therefore, researchers will compare the response of the study participants to valbenazine treatment with those from a previous reported work that resulted in the FDA approval of this medication.

DETAILED DESCRIPTION:
Tardive dyskinesia (TD) is recognized as a common and often debilitating movement disorder, associated with treatment of a variety of illnesses with dopamine receptor-blocking medications (also commonly known as antipsychotic medications. In addition to the distressing and disfiguring movements of TD, there is now also evidence of a reduced quality of life in patients with TD compared to peers with similar psychiatric disorders without TD.

When originally described, TD had been thought to be primarily associated with use of First-Generation Antipsychotics (FGA's, also known as typical antipsychotics), but there are now good studies to suggest that TD is also frequently a result of exposure to Second Generation Antipsychotics (SGA's) as well. Valbenazine, a selective vesicular monoamine transporter 2 inhibitor, is now available to treat the symptoms of TD, with a favorable efficacy and safety profile. This medication offers, for the first time, a treatment option for patients - as well as their caregivers and families - suffering with TD.

Individuals with intellectual and developmental disabilities (IDD) commonly suffer from co-occurring psychiatric and/or behavioral disorders (informally known as a "dual diagnosis"). Such individuals are commonly prescribed antipsychotic medications to treat these co-occurring disorders. Several authors have noted that antipsychotic medications have frequently been over-prescribed for individuals with IDD, often in the absence of an identified psychotic illness. Some studies have shown that up to 20-30% of adults with IDD are prescribed antipsychotic medications across a variety of residential settings.

Surrounding this frequent use of antipsychotic medications in persons with IDD, it is now well-established that persons and that having intellectual disability is a recognized risk factor for developing TD when treated with antipsychotic medications. Finally, recent research has confirmed the long-suspected belief that persons with IDD are MORE susceptible to movement disorder side effects when treated with antipsychotic medications when compared to persons without IDD.

Based on their increased exposure to antipsychotics, and increased susceptibility to movement disorders including TD, it would seem that persons with IDD who have TD are a group who could benefit most from treatment with a novel agent which can address this movement disorder.

Before TD can be treated, it must be clinically identified and formally diagnosed. Once diagnosed, patients and families must be educated on the availability of treatment options, outcomes when no treatment is undertaken, and the potential benefits (and risks) of treatment itself.

Movement disorders such as TD have been diagnosed on the basis of clinical examination, often using formal assessment tools to identify and quantify the movement abnormalities seen. One such instrument is the Abnormal Involuntary Movement Scale (AIMS). The AIMS has been used for many years as the gold standard for this purpose. In addition, there have been recent attempts to quantify the amount of improvement (change in movement intensity, and reduction in AIMS scores) that are considered clinically significant in rating improvement. Additionally, a number of authors have noted the difficulty in using the AIMS in persons with IDD who cannot cooperate fully in the examination process. For this reason, some have suggested using videotaped AIMS exams as a methodology for more accurately quantifying change. Videotaping of exams pre- and post-treatment for blind rating of improvement has been a methodology utilized in a number of recent studies of valbenazine.

In this study, 25 participants with IDD and TD will undergo valbenazine treatment for 24 weeks. The participants will be seen for a total of 5 visits: at baseline, and at follow up visits at 3 weeks, 6 weeks, 12 weeks, and 24 weeks. Consented participants will have an AIMS administered and videotaped at each visit, initially to identify and quantify TD, and subsequently to measure possible response to valbenazine. Subjects' TD response to valbenazine will also be assessed using the Clinical Global Impression of Change (CGI-C) scale (by investigator) and Caregiver Global Impression Scale (by proxy caregiver). Subjects' quality of life will be assessed with the World Health Organization Quality of Life Scale- For Persons with Disability (WHOQOL-DIS), a proxy-reported instrument designed for individuals with IDD, before and after valbenazine treatment. Participants' behavior will be assessed with the Aberrant Behavior Checklist-Irritability Subscale, before and after valbenazine treatment. Subjects' Activities of Daily Living (ADL's) will be assessed with the Waisman Activities of Daily Living Scale (W-ADL), a proxy-reported instrument designed for individuals with IDD and other disabilities, before and after valbenazine treatment. Caregiver burden will be assessed with the Zarit Burden Inventory, short version, before and after valbenazine treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IDD (IQ < 70; social/adaptive dysfunction, onset < age 22) as per DSM-5
* Clinical diagnosis of Tardive Dyskinesia (TD) per DSM-5 for at least 3 months before study inclusion (presence of movement disorder for at least 3 months, in absence of previous formal diagnosis of TD).
* Eligible to receive valbenazine according to current product labeling.
* Stable doses of all psychotropic medications for minimum of three months before study inclusion.
* Willing to remain on stable doses of all psychotropics for 24 weeks of study. If female of childbearing age, practicing acceptable form for birth control throughout study duration.
* Subject able to comply with scheduled visits and assessments.
* Consent of subject, or legally authorized representative to study protocol.

Exclusion Criteria:

* Previous treatment with a VMAT2 inhibitor (tetrabenazine, valbenazine, or deutetrabenazine).
* Treatment with any investigational drug in the 30 days prior to study entry.
* Currently taking a strong CYP3A4 inducer such as carbamazepine, phenobarbital, diphenylhydantoin, or primidone.
* Any unstable medical condition in the 60 days prior to study entry.
* Pregnant or breast-feeding.
* Inability to take study medication.
* History of neuroleptic malignant syndrome.
* History of long QTc on electrocardiogram, bundle branch block (BBB), atrioventricular block, serious cardiac arrhythmia, or heart failure.
* QTc on EKG > 450 msec (Fredericia formula) on EKG within 3 months prior to study entry.
* History of substance abuse or dependence in the 3 months prior to study entry.
* Significant risk of suicide or dangerous aggression to others at time of or 3 months prior to study entry.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in AIMS total scores of items 1-7 | Baseline and 24 weeks from start of treatment
  The Abnormal Involuntary Movement Scale (AIMS) has been used for many years as the gold standard for this purpose and the amount of improvement (change in movement intensity, and reduction in AIMS scores) have been assessed clinical significance in rating improvement. A number of authors have noted the difficulty in using the AIMS in persons with IDD who cannot cooperate fully in the examination process. For this reason, some have suggested using videotaped AIMS exams as a methodology for more accurately quantifying change. Videotaping of exams pre- and post-treatment for blind rating of improvement has been a methodology utilized in a number of recent studies of valbenazine. The minimum value of the AIMS total score of items 1-7 is 0 and the maximum value is 49. Higher total AIMS scores mean worse outcomes.

SECONDARY OUTCOMES:
Change in AIMS item 8 scores | Baseline and 24 weeks from start of treatment
  Item 8 of the AIMS represents an overall index of severity of abnormal involuntary movements. The minimum value of the AIMS total score of items 1-7 is 0 and the maximum value is 4; Higher total scores mean worse outcomes.
CGI-C | Baseline and 24 weeks from start of treatment
  Clinical Global Impression of Change (CGI-C), as the names indicates, denotes the clinician's impression of change between baseline and after the treatment in which -3 will be marked worsening, -2 moderate worsening, -1 mild worsening, 0 no change, +1 will be marked for mild improvement, +2 moderate improvement, and +3 marked improvement.
CaGI-C | Baseline and 24 weeks from start of treatment
  Caregiver Global Impression of Change (CaGI-C). This is similar to the CGI-C, except that this is the impression of the participant's caregiver, -3 will be marked worsening, -2 moderate worsening, -1 mild worsening, 0 no change, +1 will be marked for mild improvement, +2 moderate improvement, and +3 marked improvement.
Change in ABC-I score | Baseline and 24 weeks from start of treatment
  The Aberrant Behavioral Checklist, Irritability Subscale (ABC-I) is commonly used in clinical trials. It consists of 15 items, which are scored on a 4-point Likert scale of severity, ranging from "not at all a problem" to "the problem is severe in degree."
Change in W-ADL score | Baseline and 24 weeks from start of treatment
  The Waisman Activities of Daily Living (W-ADL) Scale for adolescents and adults with developmental disabilities, is a validated scale that consists of 17 items in the final version of the W-ADL pertain to the current or expected performance of the target individual at the time when the survey was given. The target adult's performance of each activity is rated on a 3-point scale (0 = "does not do at all", 1 = "does with help", 2 = "independent"), and item scores are summed to produce an overall score. Therefore, this means that the scores can range from a minimum of 0 to a maximum value of 51. Higher total W-ADL scores mean better outcomes.
Change in Zarit Burden Interview (short version) score | Baseline and 24 weeks from start of treatment
  The short version of the Zarit Burden Interview is suitable across diagnostic groups of cognitively impaired older adults, and can be used in cross-sectional, longitudinal, and intervention studies. It consists of 12 items, which are answered by a caregiver and measures the change over time, resulting from the progression of (or therapeutic effect of an intervention on) the care recipient's condition. Each item is scored on a 5-point Likert scale, with higher scores indicating greater burden, i.e., worse outcome.

OTHER OUTCOMES:
Change Simpson-Angus Scale for EPS | Baseline and 24 weeks from start of treatment
  The Simpson-Angus Scale is a tool used to assess the severity of extrapyramidal symptoms (EPS), which are side effects of antipsychotic medications. The scale consists of ten items that assess five domains: gait, arm dropping, shoulder shaking, elbow rigidity, and wrist rigidity or fixation of position. Each item is rated on a 5-point scale of severity (0 = normal; 4 = most severe; NR = not rated). The total score ranges from 0 to 40, with higher scores indicating more severe EPS outcome.
Change in Barnes Akathisia Scale | Baseline and 24 weeks from start of treatment
  The Barnes Akathisia Scale is a rating scale used to assess the severity of drug-induced akathisia (a syndrome of motor restlessness). It is the most widely used rating scale for akathisia. The scale consists of four items that rate the observable, restless movements that characterize the condition, the subjective awareness of restlessness, and any distress associated with the akathisia. The scale is scored on a 4-point scale from 0-3 and is summed yielding a total score ranging from 0 to 9. The higher the score, the more severe the akathisia, i.e., the worse the outcome.
Assessment of electrocardiogram (EKG)-derived QT/QTc intervals | Baseline and 24 weeks from start of treatment
  QTc intervals have clinical importance as a biomarker of potential drug toxicity. QTc intervals ≥ 450 ms are generally considered long, and drug-induced QTc interval prolongations ≥ 60 ms are generally considered clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ruedrich, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Trial data can be made available on reasonable request to the principal investigator and must be accompanied by detailed study proposals, a description of study objectives, and a statistical analysis plan. Access to available deidentified participant data and the trial protocol may be granted 12 months after publication.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From 12 months after publication until three years afterwards.
Access Criteria: Any request must be approved by the corresponding author and the principal investigator. Each request will be checked for compatibility with regulatory (institutional review board) requirements as well as compatibility with participant informed consent.

REFERENCES:
- [Background] Aman MG (2012) Aberrant Behavior Checklist: Current Identity and Future Developments. Clin Exp Pharmacol 2:e114. doi:10.4172/2161- 1459.1000e114
- [Background] Barnes TR. The Barnes Akathisia Rating Scale--revisited. J Psychopharmacol. 2003 Dec;17(4):365-70. doi: 10.1177/0269881103174013. PMID 14870947
- [Background] Bowring DL, Totsika V, Hastings RP, Toogood S, McMahon M. Prevalence of psychotropic medication use and association with challenging behaviour in adults with an intellectual disability. A total population study. J Intellect Disabil Res. 2017 Jun;61(6):604-617. doi: 10.1111/jir.12359. Epub 2017 Jan 16. PMID 28090687
- [Background] Correll CU, Kane JM, Citrome LL. Epidemiology, Prevention, and Assessment of Tardive Dyskinesia and Advances in Treatment. J Clin Psychiatry. 2017 Sep/Oct;78(8):1136-1147. doi: 10.4088/JCP.tv17016ah4c. PMID 29022654
- [Background] de Kuijper GM, Hoekstra PJ. Physicians' reasons not to discontinue long-term used off-label antipsychotic drugs in people with intellectual disability. J Intellect Disabil Res. 2017 Oct;61(10):899-908. doi: 10.1111/jir.12385. Epub 2017 May 30. PMID 28560761
- [Background] de Kuijper GM, Hoekstra PJ. Assessment of Drug-Associated Extrapyramidal Symptoms in People With Intellectual Disability: A Comparison of an Informant-Based Scale With Clinical Rating Scales. J Clin Psychopharmacol. 2016 Oct;36(5):508-12. doi: 10.1097/JCP.0000000000000558. PMID 27529770
- [Background] Fodstad JC, Bamburg JW, Matson JL, Mahan S, Hess JA, Neal D, Holloway J. Tardive dyskinesia and intellectual disability: an examination of demographics and topography in adults with dual diagnosis and atypical antipsychotic use. Res Dev Disabil. 2010 May-Jun;31(3):750-9. doi: 10.1016/j.ridd.2010.01.017. Epub 2010 Mar 5. PMID 20207106
- [Background] Guy W (1976). ECDEU Assessment Manual for Psychopharmacology: Revised (DHEW publication number ADM 76-338). Rockville, MD, Us Department of Health, Education and Welfare, PHS, ADAMHA, NIMH Psychopharmacology Research Branch, Division of Extramural Research Programs, 1976:534-537.
- [Background] Hauser RA, Factor SA, Marder SR, Knesevich MA, Ramirez PM, Jimenez R, Burke J, Liang GS, O'Brien CF. KINECT 3: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Trial of Valbenazine for Tardive Dyskinesia. Am J Psychiatry. 2017 May 1;174(5):476-484. doi: 10.1176/appi.ajp.2017.16091037. Epub 2017 Mar 21. PMID 28320223
- [Background] Hérbert, R., Bravo, G., & Préville, M. (2000). Reliability, validity, and reference values of the Zarit Burden Interview for assessing informal caregivers of community-dwelling older persons with dementia. Canadian Journal on Aging, 19, 494-507.
- [Background] Kane JM, Correll CU, Nierenberg AA, Caroff SN, Sajatovic M; Tardive Dyskinesia Assessment Working Group. Revisiting the Abnormal Involuntary Movement Scale: Proceedings From the Tardive Dyskinesia Assessment Workshop. J Clin Psychiatry. 2018 May/Jun;79(3):17cs11959. doi: 10.4088/JCP.17cs11959. PMID 29742330
- [Background] Maenner MJ, Smith LE, Hong J, Makuch R, Greenberg JS, Mailick MR. Evaluation of an activities of daily living scale for adolescents and adults with developmental disabilities. Disabil Health J. 2013 Jan;6(1):8-17. doi: 10.1016/j.dhjo.2012.08.005. Epub 2012 Oct 17. PMID 23260606
- [Background] Matson JL, Fodstad JC, Neal D, Dempsey T, Rivet TT. Risk factors for tardive dyskinesia in adults with intellectual disability, comorbid psychopathology, and long-term psychotropic use. Res Dev Disabil. 2010 Jan-Feb;31(1):108-16. doi: 10.1016/j.ridd.2009.08.002. Epub 2009 Aug 31. PMID 19720497
- [Background] McEvoy J, Gandhi SK, Rizio AA, Maher S, Kosinski M, Bjorner JB, Carroll B. Effect of tardive dyskinesia on quality of life in patients with bipolar disorder, major depressive disorder, and schizophrenia. Qual Life Res. 2019 Dec;28(12):3303-3312. doi: 10.1007/s11136-019-02269-8. Epub 2019 Aug 21. PMID 31435866
- [Background] Morton RO, Morton LC, Fedora R. Recognition and Treatment of Tardive Dyskinesia in Individuals with Intellectual Disability. Case Rep Psychiatry. 2020 Dec 11;2020:8886980. doi: 10.1155/2020/8886980. eCollection 2020. PMID 33414976
- [Background] Ruedrich SL. (2016). Psychopharmacology. In Hemmings C & Bouras N (eds.) Psychiatric and Behavioural Disorders in Intellectual and Developmental Disabilities, Third Edition, Cambridge University Press, Cambridge, UK, 139-150.
- [Background] Ruedrich SL (2010). Mental Illness in O'Hara J, McCarthy J, and Bouras N. (eds.) Intellectual Disability and Ill Health: A Review of the Evidence, Cambridge University Press, Cambridge UK, 165-177.
- [Background] Ruedrich SL, Diana L, Rossvanes CF, Toliver J. (2005). The abnormal involuntary movement scale (AIMS) and tardive dyskinesia in persons with developmental disability: the benefit of videotaped exams. Mental Health Aspects of Developmental Disabilities 8(3)94-99.
- [Background] Schmidt S, Power M, Green A, Lucas-Carrasco R, Eser E, Dragomirecka E, Fleck M. Self and proxy rating of quality of life in adults with intellectual disabilities: results from the DISQOL study. Res Dev Disabil. 2010 Sep-Oct;31(5):1015-26. doi: 10.1016/j.ridd.2010.04.013. Epub 2010 May 15. PMID 20478692
- [Background] Schooler NR, Kane JM. Research diagnoses for tardive dyskinesia. Arch Gen Psychiatry. 1982 Apr;39(4):486-7. doi: 10.1001/archpsyc.1982.04290040080014. No abstract available. PMID 6121550
- [Background] Sheehan R, Horsfall L, Strydom A, Osborn D, Walters K, Hassiotis A. Movement side effects of antipsychotic drugs in adults with and without intellectual disability: UK population-based cohort study. BMJ Open. 2017 Aug 3;7(8):e017406. doi: 10.1136/bmjopen-2017-017406. PMID 28775195
- [Background] Simpson GM, Angus JW. A rating scale for extrapyramidal side effects. Acta Psychiatr Scand Suppl. 1970;212:11-9. doi: 10.1111/j.1600-0447.1970.tb02066.x. No abstract available. PMID 4917967
- [Background] Solmi M, Pigato G, Kane JM, Correll CU. Clinical risk factors for the development of tardive dyskinesia. J Neurol Sci. 2018 Jun 15;389:21-27. doi: 10.1016/j.jns.2018.02.012. Epub 2018 Feb 5. PMID 29439776
- [Background] Stacy M, Sajatovic M, Kane JM, Cutler AJ, Liang GS, O'Brien CF, Correll CU. Abnormal involuntary movement scale in tardive dyskinesia: Minimal clinically important difference. Mov Disord. 2019 Aug;34(8):1203-1209. doi: 10.1002/mds.27769. Epub 2019 Jun 24. PMID 31234240
- [Background] Tsiouris JA. Pharmacotherapy for aggressive behaviours in persons with intellectual disabilities: treatment or mistreatment? J Intellect Disabil Res. 2010 Jan 1;54(1):1-16. doi: 10.1111/j.1365-2788.2009.01232.x. Epub 2009 Dec 8. PMID 20122096
- [Background] Townsend-White C, Pham AN, Vassos MV. Review: a systematic review of quality of life measures for people with intellectual disabilities and challenging behaviours. J Intellect Disabil Res. 2012 Mar;56(3):270-84. doi: 10.1111/j.1365-2788.2011.01427.x. Epub 2011 Jun 17. PMID 21679329
- [Background] Whiteney C and Evered JA (2022). The Qualitative Research Distress Protocol: A Participant-Centered Tool for Navigating Distress During Data Collection. International Journal of Qualitative Methods Volume 21:1-9.
- [Background] Woods SW, Morgenstern H, Saksa JR, Walsh BC, Sullivan MC, Money R, Hawkins KA, Gueorguieva RV, Glazer WM. Incidence of tardive dyskinesia with atypical versus conventional antipsychotic medications: a prospective cohort study. J Clin Psychiatry. 2010 Apr;71(4):463-74. doi: 10.4088/JCP.07m03890yel. Epub 2010 Feb 9. PMID 20156410
- [Background] Yu J, Yap P, Liew TM. The optimal short version of the Zarit Burden Interview for dementia caregivers: diagnostic utility and externally validated cutoffs. Aging Ment Health. 2019 Jun;23(6):706-710. doi: 10.1080/13607863.2018.1450841. Epub 2018 Mar 19. PMID 29553806